CLINICAL TRIAL: NCT06237049
Title: A Phase 1/2 Randomized Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Modified RNA COVID-19 Vaccine and a Recombinant Influenza Vaccine Administered as a Single Injection in Healthy Adults 50 Years of Age or Older
Brief Title: A Study to Learn About a Combined COVID-19 and Influenza Shot in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C5681001
Record Dates: First submitted 2024-01-30; First posted 2024-02-01 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Influenza, Human; SARS-CoV-2 Infection; COVID-19
Keywords: Grippe; Flu; Influenza Vaccine; RNA Vaccine; COVID-19; Coronavirus Vaccine; SARS-CoV-2; mRNA Vaccine
MeSH Terms: conditions — Influenza, Human; COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind (site- and sponsor-unblinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BNT162b2 (Omi XBB.1.5)/RIV and placebo (Experimental): Participants will receive a single injection combination of BNT162b2 (Omi XBB.1.5) and RIV and normal saline placebo
  Interventions: Biological: BNT162b2 (Omi XBB.1.5)/RIV; Other: Normal saline placebo
- BNT162b2 (Omi XBB.1.5) and RIV (Experimental): Participants will receive BNT162b2 (Omi XBB.1.5) and RIV
  Interventions: Biological: BNT162b2 (Omi XBB.1.5); Biological: RIV
- BNT162b2 (Omi XBB.1.5) and placebo (Active Comparator): Participants will receive BNT162b2 (Omi XBB.1.5) and normal saline placebo
  Interventions: Biological: BNT162b2 (Omi XBB.1.5); Other: Normal saline placebo
- RIV and placebo (Active Comparator): Participants will receive RIV and normal saline placebo
  Interventions: Biological: RIV; Other: Normal saline placebo

INTERVENTIONS:
Biological: BNT162b2 (Omi XBB.1.5)/RIV — Combination of BNT162b2 (Omi XBB.1.5) and RIV
  Arms: BNT162b2 (Omi XBB.1.5)/RIV and placebo
Biological: BNT162b2 (Omi XBB.1.5) — Licensed COVID-19 vaccine
  Arms: BNT162b2 (Omi XBB.1.5) and RIV; BNT162b2 (Omi XBB.1.5) and placebo
Biological: RIV — Licensed recombinant influenza vaccine
  Arms: BNT162b2 (Omi XBB.1.5) and RIV; RIV and placebo
Other: Normal saline placebo — Normal saline (solution for injection)
  Arms: BNT162b2 (Omi XBB.1.5) and placebo; BNT162b2 (Omi XBB.1.5)/RIV and placebo; RIV and placebo

SUMMARY:
The purpose of this clinical trial is to see if combining a licensed COVID-19 vaccine and a licensed influenza vaccine into a single shot is safe and can help produce antibodies to defend the body against both SARS-CoV-2 (the virus that causes COVID-19) and influenza. Participants enrolled in this trial will be healthy adults, 50 years of age or older.

DETAILED DESCRIPTION:
This is a Phase 1/2 study to evaluate the safety, tolerability, and immunogenicity of licensed BNT162b2 (Omi XBB.1.5) and recombinant influenza vaccine (RIV) administered together as a single injection (referred to as BNT162b2 [Omi XBB.1.5]/RIV) in healthy adults 50 years of age or older.

The safety, tolerability, and immunogenicity of BNT162b2 (OmiXBB1.5)/RIV administered as a single injection will be compared to BNT162b2 (Omi XBB.1.5) and RIV administered simultaneously as 2 separate injections (coadministered), and to BNT162b2 (Omi XBB.1.5) or RIV when administered alone.

Across Phases 1 and 2, approximately 640 participants in total will be randomized with an equal randomization ratio to 1 of 4 vaccine groups and stratified by age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 50 years or older at Visit 1 (Day 1).
* Participants who are willing and able to comply with all scheduled visits, the investigational plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* Capable of giving signed informed consent as described in the protocol, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in the protocol.

Exclusion Criteria:

* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Known infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
* History of severe adverse reaction associated with any vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study interventions.
* Participants with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to systemic or cutaneous lupus erythematosus, autoimmune arthritis/rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, idiopathic thrombocytopenia purpura, glomerulonephritis, autoimmune thyroiditis, temporal arteritis, psoriasis, and/or insulin-dependent diabetes mellitus.
* Immunocompromised individuals with known or suspected immunodeficiency, determined by history and/or laboratory/physical examination.
* Current heart disease, uncontrolled hypertension, or a prior history of myocarditis or pericarditis.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant, plan to become pregnant during the study, or are breastfeeding.
* Prior history of ischemic stroke or transient ischemic attack.
* Prior history of Guillain-Barré syndrome (GBS).
* Participants with a calculated BMI of ≥35.
* Receipt of chronic medications with known systemic immunosuppressant effects (including cytotoxic agents or systemic corticosteroids), or radiotherapy, within 60 days before enrollment through conclusion of the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies used for the treatment or prevention of COVID 19 or those that are considered immunosuppressive, from 90 days before study intervention administration, or planned receipt throughout the study.
* Vaccination with any investigational or licensed influenza vaccine within 6 months (180 days) before study intervention administration, or ongoing receipt of chronic antiviral therapy with activity against influenza.
* Vaccination with any investigational or licensed COVID-19 vaccine within 6 months (180 days) before study intervention administration.
* Participation in other studies involving administration of an investigational product within 28 days prior to, and/or during, participation in this study.
* Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction that in the opinion of the investigator might interfere with the study conduct or completion.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (30):
  - Orange County Research Center, Lake Forest, California
  - Orange County Research Center, Tustin, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research Consulting, Milford, Connecticut
  - GW Medical Faculty Associates, Washington D.C., District of Columbia
  - GW Vaccine Research Unit, Washington D.C., District of Columbia
  - JEM Research Institute, Atlantis, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Optimal Research, Melbourne, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Optimal Research, Peoria, Illinois
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO, Springfield, Missouri
  - Bio-Kinetic Clinical Applications, LLD dba QPS-MO, Springfield, Missouri
  - Bio-Kinetic Clinical Applications LLC DBA QPS-MO(Patient Screening Center), Springfield, Missouri
  - Las Vegas Clinical Trials, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - ActivMed Practices & Research, LLC., Portsmouth, New Hampshire
  - Rochester Clinical Research, LLC, Rochester, New York
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Clinical Research Associates Inc, Nashville, Tennessee
  - DM Clinical Research- Cyfair, Houston, Texas
  - DM Clinical Research - Bellaire, Houston, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - DM Clinical Research - MDC, Tomball, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5681001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive licensed Pfizer-BioNTech COVID-19 vaccine (BNT162b2 [Omi XBB.1.5]) 30 microgram (mcg) and recombinant influenza virus (RIV) vaccine 180 mcg together as a single injection or as 2 separate injections co-administered or BNT162b2 (Omi XBB.1.5) 30 mcg administered alone or RIV 180 mcg administered alone.
Groups:
- Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo: Participants were randomized to receive BNT162b2 (Omi XBB.1.5)/RIV together as a single intramuscular (IM) injection in the left deltoid and normal saline placebo IM injection in the right deltoid on Day 1.
- Group 2: BNT162b2 (Omi XBB.1.5) + RIV: Participants were randomized to receive BNT162b2 (Omi XBB.1.5) IM injection in the left deltoid and RIV IM injection in the right deltoid on Day 1.
- Group 3: BNT162b2 (Omi XBB.1.5) + Placebo: Participants were randomized to receive BNT162b2 (Omi XBB.1.5) IM injection in the left deltoid and normal saline placebo IM injection in the right deltoid on Day 1.
- Group 4: RIV + Placebo: Participants were randomized to receive RIV IM injection in the left deltoid and normal saline placebo IM injection in the right deltoid on Day 1.
Period: Overall Study
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 3: BNT162b2 (Omi XBB.1.5) + Placebo | Group 4: RIV + Placebo
Started | 160 | 163 | 160 | 161
Vaccinated | 160 | 161 | 160 | 160
Completed | 145 | 155 | 151 | 151
Not Completed | 15 | 8 | 9 | 10
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 11 | 5 | 8 | 8
Not completed — Protocol Violation | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) consisted of all participants who received at least 1 dose of the study intervention.
Groups:
- Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo: Participants were randomized to receive BNT162b2 (Omi XBB.1.5)/RIV together as a single IM injection in the left deltoid and normal saline placebo IM injection in the right deltoid on Day 1.
- Total: Total of all reporting groups
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 3: BNT162b2 (Omi XBB.1.5) + Placebo | Group 4: RIV + Placebo | Total
Number analyzed (Participants) | 160 | 161 | 160 | 160 | 641
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (8.40) | 63.9 (9.06) | 62.9 (7.73) | 63.9 (7.66) | 63.7 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 92 | 100 | 83 | 362
  Male | 73 | 69 | 60 | 77 | 279
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 28 | 29 | 21 | 106
  Not Hispanic or Latino | 132 | 133 | 131 | 137 | 533
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 1 | 4
  Asian | 5 | 6 | 3 | 6 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2 | 4
  Black or African American | 37 | 38 | 30 | 30 | 135
  White | 117 | 111 | 124 | 117 | 469
  More than one race | 0 | 2 | 2 | 2 | 6
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Reported Any Local Reaction up to 7 Days Following Vaccination
Description: Local reactions included redness, swelling and pain at injection site, recorded by participants in an electronic diary (e-diary). Severity of all local reactions were evaluated as mild, moderate, severe or potentially life-threatening. In this outcome measure local reactions with any severity were reported for each left arm's deltoid and right arm's deltoid of each vaccine Group 1, 2, 3 and 4.
Time Frame: Day 1 to Day 7 following Vaccination on Day 1
Population: SAS consisted of all participants who received at least 1 dose of the study intervention. As planned, results of this outcome measure are reported for vaccination in each arm (left and right deltoid- as separate reporting arm) of each vaccine group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Group 1, BNT162b2/RIV + Placebo: BNT162b2/RIV: Participants received BNT162b2/RIV as a single IM injection in the left deltoid.
- Group 1, BNT162b2/RIV + Placebo: Placebo; Group 3, BNT162b2 + Placebo: Placebo; Group 4, RIV + Placebo: Placebo: Participants received normal saline placebo IM injection in the right deltoid.
- Group 2, BNT162b2 + RIV: BNT162b2; Group 3, BNT162b2 + Placebo: BNT162b2: Participants received BNT162b2 (Omi XBB.1.5) IM injection in the left deltoid.
- Group 2, BNT162b2 + RIV: RIV: Participants received RIV IM injection in the right deltoid.
- Group 4, RIV + Placebo: RIV: Participants received RIV IM injection in the left deltoid.
Arm/Group | Group 1, BNT162b2/RIV + Placebo: BNT162b2/RIV | Group 1, BNT162b2/RIV + Placebo: Placebo | Group 2, BNT162b2 + RIV: BNT162b2 | Group 2, BNT162b2 + RIV: RIV | Group 3, BNT162b2 + Placebo: BNT162b2 | Group 3, BNT162b2 + Placebo: Placebo | Group 4, RIV + Placebo: RIV | Group 4, RIV + Placebo: Placebo
Number analyzed (Participants) | 160 | 160 | 161 | 161 | 160 | 160 | 160 | 160
Percentage of participants
  Pain at injection site | 56.3 [48.2 to 64.1] | 11.9 [7.3 to 17.9] | 59.0 [51.0 to 66.7] | 38.5 [31.0 to 46.5] | 62.5 [54.5 to 70.0] | 9.4 [5.3 to 15.0] | 36.9 [29.4 to 44.9] | 8.1 [4.4 to 13.5]
  Redness | 8.8 [4.9 to 14.2] | 1.3 [0.2 to 4.4] | 5.0 [2.2 to 9.6] | 3.1 [1.0 to 7.1] | 5.0 [2.2 to 9.6] | 0.6 [0.0 to 3.4] | 6.3 [3.0 to 11.2] | 0.6 [0.0 to 3.4]
  Swelling | 9.4 [5.3 to 15.0] | 1.3 [0.2 to 4.4] | 6.2 [3.0 to 11.1] | 3.1 [1.0 to 7.1] | 5.6 [2.6 to 10.4] | 0.6 [0.0 to 3.4] | 5.0 [2.2 to 9.6] | 0.6 [0.0 to 3.4]

2. Primary Outcome: Percentage of Participants Who Reported Any Systemic Events up to 7 Days Following Vaccination
Description: Systemic events: fever, fatigue, headache, vomiting, diarrhea, chills, new/worsened muscle pain, new/worsened joint pain were recorded by participants in e-diary. Severity of all systemic events were evaluated as mild, moderate, severe or potentially life-threatening. In this outcome measure systemic events with any severity were reported.
Time Frame: Day 1 to Day 7 following Vaccination on Day 1
Population: SAS consisted of all participants who received at least 1 dose of the study intervention. Data is presented for each vaccine group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 3: BNT162b2 (Omi XBB.1.5) + Placebo | Group 4: RIV + Placebo
Number analyzed (Participants) | 160 | 161 | 160 | 160
Percentage of participants
  Fever | 1.9 [0.4 to 5.4] | 6.2 [3.0 to 11.1] | 6.3 [3.0 to 11.2] | 0 [0.0 to 2.3]
  Fatigue | 36.3 [28.8 to 44.2] | 39.1 [31.5 to 47.1] | 40.6 [32.9 to 48.7] | 33.1 [25.9 to 41.0]
  Headache | 24.4 [17.9 to 31.8] | 31.1 [24.0 to 38.8] | 26.9 [20.2 to 34.4] | 16.9 [11.4 to 23.6]
  Vomiting | 0 [0.0 to 2.3] | 3.1 [1.0 to 7.1] | 1.9 [0.4 to 5.4] | 0 [0.0 to 2.3]
  Diarrhea | 8.1 [4.4 to 13.5] | 11.2 [6.8 to 17.1] | 11.3 [6.8 to 17.2] | 7.5 [3.9 to 12.7]
  Chills | 8.8 [4.9 to 14.2] | 14.9 [9.8 to 21.4] | 15.0 [9.9 to 21.5] | 6.9 [3.5 to 12.0]
  New or worsened muscle pain | 13.1 [8.3 to 19.4] | 22.4 [16.2 to 29.6] | 15.0 [9.9 to 21.5] | 8.1 [4.4 to 13.5]
  New or worsened joint pain | 7.5 [3.9 to 12.7] | 13.7 [8.8 to 20.0] | 10.0 [5.8 to 15.7] | 4.4 [1.8 to 8.8]

3. Primary Outcome: Percentage of Participants Who Reported Any Adverse Events (AEs) From Vaccination Through 4 Weeks After Vaccination
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Events collected by systematic assessment (local reactions and systemic events) were excluded from evaluation.
Time Frame: From Vaccination on Day 1 through 4 weeks after Vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 3: BNT162b2 (Omi XBB.1.5) + Placebo | Group 4: RIV + Placebo
Number analyzed (Participants) | 160 | 161 | 160 | 160
Percentage of participants | 4.4 [1.8 to 8.8] | 3.7 [1.4 to 7.9] | 5.6 [2.6 to 10.4] | 5.6 [2.6 to 10.4]

4. Primary Outcome: Percentage of Participants Who Reported Any Serious Adverse Events (SAEs) From Vaccination Through 6 Months After Vaccination
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect and other important medical events per protocol of the study. Events collected by systematic assessment (local reactions and systemic events) were excluded from evaluation.
Time Frame: From Vaccination on Day 1 through 6 months after Vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 3: BNT162b2 (Omi XBB.1.5) + Placebo | Group 4: RIV + Placebo
Number analyzed (Participants) | 160 | 161 | 160 | 160
Percentage of participants | 1.9 [0.4 to 5.4] | 0.6 [0.0 to 3.4] | 0 [0.0 to 2.3] | 1.9 [0.4 to 5.4]

5. Primary Outcome: Geometric Mean Titers (GMTs) of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Omicron (XBB.1.5)-Neutralizing Titers Before Vaccination
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). As planned, outcome measure evaluated GMTs of SARS-CoV-2 Omicron (XBB.1.5), hence results are reported only for those reporting groups where BNT162b2 (Omi XBB.1.5) was administered. Data was not collected and not reported for reporting group "Group 4: RIV + Placebo", where BNT162b2 (Omi XBB.1.5) was not administered.
Time Frame: Before Vaccination on Day 1
Population: Evaluable immunogenicity population (EIP) included all eligible participants who received study intervention, had at least 1 valid and determinate immunogenicity result from the blood sample collected within 27 to 42 days after vaccination, and had no other important protocol deviations as determined by the clinician. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 3: BNT162b2 (Omi XBB.1.5) + Placebo
Number analyzed (Participants) | 151 | 157 | 154
Titer | 311.2 [236.2 to 409.9] | 285.4 [220.4 to 369.5] | 338.5 [256.9 to 446.0]

6. Primary Outcome: GMTs of SARS-CoV-2 Omicron (XBB.1.5)-Neutralizing Titers at 4 Weeks After Vaccination
Description: as for outcome 5
Time Frame: At 4 weeks after Vaccination on Day 1
Population: EIP included all eligible participants who received study intervention, had at least 1 valid and determinate immunogenicity result from the blood sample collected within 27 to 42 days after vaccination, and had no other important protocol deviations as determined by the clinician. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 3: BNT162b2 (Omi XBB.1.5) + Placebo
Number analyzed (Participants) | 151 | 158 | 152
Titer | 2162.4 [1719.6 to 2719.4] | 2581.3 [2076.2 to 3209.5] | 3644.7 [2853.7 to 4654.8]

7. Primary Outcome: Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Omicron (XBB.1.5)-Neutralizing Titers From Before Vaccination to 4 Weeks After Vaccination
Description: GMFR was the ratio of the geometric mean titre values 4 weeks after vaccination to before vaccination. GMFRs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). As planned, outcome measure evaluated GMTs of SARS-CoV-2 Omicron (XBB.1.5), hence results are reported only for those reporting groups where BNT162b2 (Omi XBB.1.5) was administered. Data was not collected and not reported for reporting group "Group 4: RIV + Placebo", where BNT162b2 (Omi XBB.1.5) was not administered.
Time Frame: From before Vaccination on Day 1 to 4 weeks after Vaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 3: BNT162b2 (Omi XBB.1.5) + Placebo
Number analyzed (Participants) | 149 | 157 | 152
Ratio | 6.1 [4.7 to 7.9] | 8.0 [6.3 to 10.1] | 9.4 [7.2 to 12.3]

8. Primary Outcome: Percentages of Participants With Seroresponse to SARS-CoV-2 Omicron (XBB.1.5) at 4 Weeks After Vaccination
Description: Seroresponse was defined as achieving a >=4-fold rise from baseline (before the study vaccination). If the baseline measurement was below the lower limit of quantification (LLOQ), the postvaccination measure of >=4*LLOQ is considered a seroresponse. Exact 2-sided CI, based on the Clopper and Pearson method. As planned, outcome measure evaluated GMTs of SARS-CoV-2 Omicron (XBB.1.5), hence results are reported only for those reporting groups where BNT162b2 (Omi XBB.1.5) was administered. Data was not collected and not reported for reporting group "Group 4: RIV + Placebo", where BNT162b2 (Omi XBB.1.5) was not administered.
Time Frame: At 4 weeks after Vaccination on Day 1
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 3: BNT162b2 (Omi XBB.1.5) + Placebo
Number analyzed (Participants) | 149 | 157 | 152
Percentage of participants | 53.7 [45.3 to 61.9] | 60.5 [52.4 to 68.2] | 63.8 [55.6 to 71.4]

9. Primary Outcome: GMTs of Strain Specific Hemagglutinin Inhibition Assay (HAI) Titers Before Vaccination
Description: GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). The 4 virus strains which were evaluated and reported in this outcome measure were A/Victoria/4897/2022 (H1N1) HAI, A/Darwin/9/2021 (H3N2) HAI, B/Michigan/1/2021 HAI and B/Phuket/3073/2013 HAI. As planned, outcome measure evaluated GMTs of strain specific HAI, hence results are reported only for those reporting groups where RIV was administered. Data was not collected and not reported for reporting group "Group 3: BNT162b2 (Omi XBB.1.5) + Placebo", where RIV was not administered.
Time Frame: Before Vaccination on Day 1
Population: EIP included all eligible participants who received study intervention, had at least 1 valid and determinate immunogenicity result from the blood sample collected within 27 to 42 days after vaccination, and had no other important protocol deviations as determined by the clinician.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 4: RIV + Placebo
Number analyzed (Participants) | 153 | 158 | 155
Titer
  A/Victoria/4897/ 2022 (H1N1) HAI | 43.8 [33.9 to 56.5] | 60.7 [47.7 to 77.1] | 62.6 [49.0 to 79.8]
  A/Darwin/9/ 2021 (H3N2) HAI | 34.8 [26.8 to 45.1] | 42.3 [32.7 to 54.9] | 44.3 [33.8 to 58.1]
  B/Michigan/1/ 2021 HAI | 105.9 [82.4 to 136.2] | 101.8 [81.4 to 127.4] | 114.9 [92.0 to 143.6]
  B/Phuket/3073/ 2013 HAI | 186.6 [151.8 to 229.5] | 218.5 [181.3 to 263.2] | 228.8 [185.9 to 281.7]

10. Primary Outcome: GMTs of Strain Specific Hemagglutinin Inhibition Assay (HAI) Titers at 4 Weeks After Vaccination
Description: as for outcome 9
Time Frame: At 4 weeks after Vaccination on Day 1
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 4: RIV + Placebo
Number analyzed (Participants) | 153 | 158 | 155
Titer
  A/Victoria/4897/ 2022 (H1N1) HAI | 324.4 [250.4 to 420.2] | 374.7 [299.4 to 469.1] | 389.6 [309.4 to 490.5]
  A/Darwin/9/ 2021 (H3N2) HAI | 397.7 [310.4 to 509.7] | 489.7 [393.9 to 608.9] | 557.2 [440.8 to 704.2]
  B/Michigan/1/ 2021 HAI | 464.0 [384.5 to 559.9] | 427.5 [360.0 to 507.6] | 496.0 [408.6 to 602.1]
  B/Phuket/3073/ 2013 HAI | 669.7 [568.4 to 789.0] | 769.5 [658.9 to 898.7] | 775.7 [656.1 to 917.1]

11. Primary Outcome: GMFR of Strain Specific HAI Titers From Before Vaccination to 4 Weeks After Vaccination
Description: GMFR was the ratio of the geometric mean titre values 4 weeks after vaccination to before vaccination. GMFRs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). The 4 virus strains which were evaluated and reported in this outcome measure were A/Victoria/4897/2022 (H1N1) HAI, A/Darwin/9/2021 (H3N2) HAI, B/Michigan/1/2021 HAI and B/Phuket/3073/2013 HAI. As planned, outcome measure evaluated GMFRs of strain specific HAI, hence results are reported only for those reporting groups where RIV was administered. Data was not collected and not reported for reporting group "Group 3: BNT162b2 (Omi XBB.1.5) + Placebo", where RIV was not administered.
Time Frame: From before Vaccination to 4 weeks after Vaccination on Day 1
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 4: RIV + Placebo
Number analyzed (Participants) | 153 | 158 | 155
Ratio
  A/Victoria/4897/ 2022 (H1N1) HAI | 6.6 [5.2 to 8.5] | 5.7 [4.5 to 7.2] | 5.7 [4.5 to 7.2]
  A/Darwin/9/ 2021 (H3N2) HAI | 9.9 [7.7 to 12.6] | 10.1 [8.0 to 12.8] | 11.0 [8.5 to 14.3]
  B/Michigan/1/ 2021 HAI | 4.3 [3.5 to 5.3] | 4.1 [3.4 to 5.0] | 4.2 [3.3 to 5.4]
  B/Phuket/3073/ 2013 HAI | 3.6 [2.9 to 4.4] | 3.5 [2.9 to 4.2] | 3.4 [2.8 to 4.1]

12. Primary Outcome: Percentages of Participants Achieving HAI Seroconversion at 4 Weeks After Vaccination
Description: Seroconversion was defined as an HAI titer <1:10 prior to vaccination and >=1:40 at the time point of interest, or an HAI titer of >=1:10 prior to vaccination with a minimum 4-fold rise at the time point of interest. Exact 2-sided CI, based on the Clopper and Pearson method. The 4 virus strains which were evaluated and reported in this outcome measure were A/Victoria/4897/2022 (H1N1) HAI, A/Darwin/9/2021 (H3N2) HAI, B/Michigan/1/2021 HAI and B/Phuket/3073/2013 HAI. As planned, outcome measure evaluated seroconversion of strain specific HAI, hence results are reported only for those reporting groups where RIV was administered. Data was not collected and not reported for reporting group "Group 3: BNT162b2 (Omi XBB.1.5) + Placebo", where RIV was not administered.
Time Frame: At 4 weeks after Vaccination on Day 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 4: RIV + Placebo
Number analyzed (Participants) | 153 | 158 | 155
Percentage of participants
  A/Victoria/4897/ 2022 (H1N1) HAI | 62.7 [54.6 to 70.4] | 67.7 [59.8 to 74.9] | 61.3 [53.1 to 69.0]
  A/Darwin/9/2021 (H3N2) | 76.5 [68.9 to 82.9] | 79.1 [71.9 to 85.2] | 76.1 [68.6 to 82.6]
  B/Michigan/1/2021 | 54.9 [46.7 to 62.9] | 53.2 [45.1 to 61.1] | 51.0 [42.8 to 59.1]
  B/Phuket/3073/2013 | 49.7 [41.5 to 57.9] | 53.8 [45.7 to 61.8] | 46.5 [38.4 to 54.6]

13. Primary Outcome: Percentages of Participants With HAI Titers >= 1:40 Before Vaccination
Description: Percentages of participants with HAI titers >= 1:40 before vaccination along with the associated 2-sided 95% CIs, was provided for each vaccine group in this outcome measure. Exact 2-sided CI, based on the Clopper and Pearson method. The 4 virus strains which were evaluated and reported in this outcome measure were A/Victoria/4897/2022 (H1N1) HAI, A/Darwin/9/2021 (H3N2) HAI, B/Michigan/1/2021 HAI and B/Phuket/3073/2013 HAI. As planned, outcome measure evaluated of strain specific HAI, hence results are reported only for those reporting groups where RIV was administered. Data was not collected and not reported for reporting group "Group 3: BNT162b2 (Omi XBB.1.5) + Placebo", where RIV was not administered.
Time Frame: Before Vaccination on Day 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 4: RIV + Placebo
Number analyzed (Participants) | 153 | 158 | 155
Percentage of participants
  A/Victoria/4897/ 2022 (H1N1) HAI | 55.6 [47.3 to 63.6] | 69.6 [61.8 to 76.7] | 70.3 [62.5 to 77.4]
  A/Darwin/9/2021 (H3N2) | 49.7 [41.5 to 57.9] | 57.6 [49.5 to 65.4] | 54.8 [46.7 to 62.8]
  B/Michigan/1/2021 | 74.5 [66.8 to 81.2] | 81.6 [74.7 to 87.3] | 81.3 [74.2 to 87.1]
  B/Phuket/3073/2013 | 89.5 [83.6 to 93.9] | 94.3 [89.5 to 97.4] | 93.5 [88.5 to 96.9]

14. Primary Outcome: Percentages of Participants With HAI Titers >= 1:40 at 4 Weeks After Vaccination
Description: Percentages of participants with HAI titers >= 1:40 at 4 weeks after vaccination along with the associated 2-sided 95% CIs, was provided for each vaccine group in this outcome measure. Exact 2-sided CI, based on the Clopper and Pearson method. The 4 virus strains which were evaluated and reported in this outcome measure were A/Victoria/4897/2022 (H1N1) HAI, A/Darwin/9/2021 (H3N2) HAI, B/Michigan/1/2021 HAI and B/Phuket/3073/2013 HAI. As outcome measure evaluated of strain specific HAI, hence results are reported only for those reporting groups where RIV was administered. Data was not collected and not reported for reporting group "Group 3: BNT162b2 (Omi XBB.1.5) + Placebo", where RIV was not administered.
Time Frame: At 4 Weeks after Vaccination on Day 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 4: RIV + Placebo
Number analyzed (Participants) | 153 | 158 | 155
Percentage of participants
  A/Victoria/4897/ 2022 (H1N1) HAI | 90.8 [85.1 to 94.9] | 95.6 [91.1 to 98.2] | 96.8 [92.6 to 98.9]
  A/Darwin/9/2021 (H3N2) | 95.4 [90.8 to 98.1] | 97.5 [93.6 to 99.3] | 96.1 [91.8 to 98.6]
  B/Michigan/1/2021 | 98.0 [94.4 to 99.6] | 100.0 [97.7 to 100.0] | 99.4 [96.5 to 100.0]
  B/Phuket/3073/2013 | 99.3 [96.4 to 100.0] | 100.0 [97.7 to 100.0] | 100.0 [97.6 to 100.0]

ADVERSE EVENTS:
Time Frame: AEs by systematic assessment: Day 1 up to 7 Days following Vaccination; AEs by Non-systematic assessment: a) Serious AEs- Day 1 of Vaccination up to 6 months of follow-up after Vaccination, b) Other AEs- Day 1 of Vaccination up to 4 weeks of follow-up after Vaccination; All-cause mortality: Day 1 of Vaccination up to 6 months of follow-up after Vaccination
Description: Same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Safety population consisted of all randomized participants who received study intervention. Data is reported for each vaccine Group.
Groups:
- Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo: Participants were randomized to receive BNT162b2 (Omi XBB.1.5)//RIV together as a single IM injection in the left deltoid and normal saline placebo IM injection in the right deltoid on Day 1.
Arm/Group | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo | Group 2: BNT162b2 (Omi XBB.1.5) + RIV | Group 3: BNT162b2 (Omi XBB.1.5) + Placebo | Group 4: RIV + Placebo
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/161 | 0/160 | 1/160
Serious Adverse Events (participants affected / at risk) | 3/160 | 1/161 | 0/160 | 3/160
Other Adverse Events (participants affected / at risk) | 114/160 | 117/161 | 115/160 | 88/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo (N=160) | Group 2: BNT162b2 (Omi XBB.1.5) + RIV (N=161) | Group 3: BNT162b2 (Omi XBB.1.5) + Placebo (N=160) | Group 4: RIV + Placebo (N=160)
Death (General disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: BNT162b2 (Omi XBB.1.5)/ RIV + Placebo (N=160) | Group 2: BNT162b2 (Omi XBB.1.5) + RIV (N=161) | Group 3: BNT162b2 (Omi XBB.1.5) + Placebo (N=160) | Group 4: RIV + Placebo (N=160)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0
Vessel puncture site haemorrhage (General disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Norovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Chills (CHILLS) (General disorders) | 14 | 24 | 24 | 11
Fatigue (FATIGUE) (General disorders) | 58 | 63 | 65 | 53
Injection site erythema (REDNESS) left deltoid (General disorders) | 14 | 8 | 8 | 10
Injection site erythema (REDNESS) right deltoid (General disorders) | 2 | 5 | 1 | 1
Injection site pain (PAIN AT THE INJECTION SITE) left deltoid (General disorders) | 90 | 95 | 100 | 59
Injection site pain (PAIN AT THE INJECTION SITE) right deltoid (General disorders) | 19 | 62 | 15 | 13
Injection site swelling (SWELLING) left deltoid (General disorders) | 15 | 10 | 9 | 8
Injection site swelling (SWELLING) right deltoid (General disorders) | 2 | 5 | 1 | 1
Pyrexia (FEVER) (General disorders) | 3 | 10 | 10 | 0
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 13 | 18 | 18 | 12
Vomiting (VOMITING) (Gastrointestinal disorders) | 0 | 5 | 3 | 0
Arthralgia (NEW OR WORSENED JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 12 | 22 | 16 | 7
Myalgia (NEW OR WORSENED MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 21 | 36 | 24 | 13
Headache (HEADACHE) (Nervous system disorders) | 39 | 50 | 43 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT06237049/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT06237049/SAP_001.pdf